CLINICAL TRIAL: NCT06439875
Title: Effects of the Association of L-arginine and Liposomal Vitamin C on Fatigue in COPD Patients With Chronic Respiratory Failure After Rehabilitation Intervention
Brief Title: Effects of L-arginine and Liposomial Vitamin C on Severe Copd Patients Undergoing Pulmonary Rehabilitation.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Collaborators: Azienda Ospedaliera dei Colli (Other); Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTSM109-23
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Respiratory Failure
Keywords: COPD; pulmonary rehabilitation; L-arginine; fatigue; respiratory failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Insufficiency; Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine (arm 1) (Experimental): Participants in this arm of the study will have an oral supplementation of l-arginine and liposomial vitamin C on a daily basis for 28 days.
  Interventions: Dietary Supplement: effect of L-arginine and liposomial vitamin C on pulmonary rehabilitation
- Placebo (arm 2) (Placebo Comparator): This arm will be given a placebo comparator on a daily basis for 28 days.
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: effect of L-arginine and liposomial vitamin C on pulmonary rehabilitation — Patients with a certified diagnosis of COPD and chronic respiratory failure will be randomized in a 1:1 ratio into the interventional arm or the placebo controller arm. All patients will undergo multidisciplinary intensive pulmonary rehabilitation for 28 days. The patients in the interventional group will receive a twice-daily oral supplementation with either a combination of 1.66 g l-arginine plus 500 mg liposomal vitamin C
  Arms: L-arginine (arm 1)
Other: placebo — Patients in this arm will undergo multidisciplinary intensive pulmonary rehabilitation without any dietary supplementation.
  Arms: Placebo (arm 2)

SUMMARY:
The hypothesis that is being tested is that the supplementation of L-arginine plus Vitamin C to multidisciplinary pulmonary rehabilitation (PR) in patients with a previous diagnosis of chronic obstructive pulmonary disease (COPD) and chronic respiratory failure can have a favorable influence on fatigue and on clinical indicators related to endothelial function, potentially mitigating the cardiovascular (CV) disease burden in this clinical context.

DETAILED DESCRIPTION:
The primary objective of this project is to assess the effects of L-arginine plus Vitamin C supplementation on the physical outcomes in a group of COPD patients with chronic respiratory failure who underwent a 28-day PR program.

Eligible participants will be randomized using a random number generator in a 1:1 ratio to receive a twice-daily oral supplementation with either a combination of 1.66 g l-arginine plus 500 mg liposomal vitamin C (Bioarginina® C, Farmaceutici Damor, Naples, Italy) or a placebo for 28 days. Vials containing the active supplement or the placebo will be supplied by Farmaceutici Damor and will be made indistinguishable in appearance. All patients will undergo an intensive multidisciplinary PR program based on endurance and strength training. The main outcome of the study is the fatigue severity scale (FSS) total score after rehabilitation. Secondary outcomes include: 6-minute walking distance, forced expiratory volume in the first second (FEV1), COPD assessment test (CAT) score, endothelial function assessed through flow-mediated dilation (FMD), and muscular strength assessed through handgrip measurement.

Anthropometric, clinical, and functional characteristics of the study participants will be reported as mean ± standard deviation (SD) or median (interquartile range, IQR) for continuous variables and as absolute values (percentages) for categorical variables. Changes from baseline for continuous variables will be expressed as deltas (values at 28 days minus the values at baseline), and differences between the interventional groups will be evaluated using the Student's t-test for normally distributed variables or the Mann-Whitney U test for skewed variables.

ELIGIBILITY:
Inclusion criteria:

* COPD patients of both sexes complicated by respiratory failure (PaO2 inferior to 60 mmHg while breathing room air)
* aged between 40 and 90 years selected from the inpatient/outpatient population admitted to perform a PR program in 12 Italian rehabilitation hospitals.

Exclusion criteria:

* consuming any ergogenic supplement in the last 2 months;
* severe acute exacerbations in the 3 months before enrolment;
* clinical instability (pH inferior to 7.35, hemodynamic instability, tachypnea at rest);
* lung restrictive diseases;
* primitive pulmonary hypertension;
* recent lung thromboembolic events;
* orthopaedic clinical conditions interfering with exercise;
* coronary heart disease;
* cardiac failure with reduced ejection fraction;
* major cardiac arrhythmias;
* neuromuscular diseases;
* mini mental state examination (MMSE) <24;
* any prior or current medical problem that would limit the subject participation

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale | at baseline and after 28 days of intensive pulmonary rehabilitation
  The Fatigue Severity Scale (FSS) is a 9-item scale that measures the severity of fatigue and how much it affects the person's activities and lifestyle in patients with a variety of disorders. The items are scored on a 7 point scale with 1=strongly disagree and 7=strongly agree. The minimum score=9 and maximum score possible=63. Higher the score=greater fatigue severity. More common way of scoring: mean of all the scores with minimum score being 1 and maximum score being 7. Mean (SD) FSS scores for healthy individuals; 2.3 (0.7). Cut-off score of 4 or more considered indicative of problematic fatigue.

SECONDARY OUTCOMES:
Six minute walking test (6MWT) | at baseline and after 28 days of intensive pulmonary rehabilitation
  The six minute walking test (6MWT) is a strong predictor of survival and outcome in PR. The patient is asked to walk on a flat surface for six minutes. The total distance walked, peripheral saturation, heart rate, dyspnea and muscular fatigue are assessed before starting the test and at the end. The distance walked varies with age and might be affected by non-respiratory diseases such as musculoscheletal and cardiovascular diseases. A distance walked inferior to the 80% of the theoretical distance is considered to be abnormal, as well as the presence of desaturations defined as a peripheral oxygen saturation < 90%. Dyspnea and fatigue are assessed through the modified Borg's scale, which ranges from 0 (= no symptom) to 10 (the most intense sensation imaginable).
Sit to stand test (STST) | at baseline and after 28 days of intensive pulmonary rehabilitation
  The participant is coached to perform as many full stands as possible within 30 seconds, starting from and returning to a complete sitting position.
  It is possible to assess a wide variety of ability levels with scores ranging from 0 for those who can not complete one stand to a score greater than 20 for more fit individuals.
COPD Assessment Test (CAT) | at baseline and after 28 days of intensive pulmonary rehabilitation
  CAT is designed to measure the impact of COPD on a person's life, and how this changes over time.
  CAT explores eight different domains, and for each one the participant may indicate a score ranging from 0 to 5. A score of 0 means that there is no impairment in that area. A score of 5 means severe impairment.The overall score will therefore range from 0 to 40. Higher scores indicate that COPD has a greater impact on the patient's overall health and well-being.
Medical Research Council (MRC) for dyspnea test | at baseline and after 28 days of intensive pulmonary rehabilitation
  MRC uses to assess the degree of baseline functional disability due to dyspnoea. It ranges from 0 to 4. A value = 0 indicates no significant dyspnea. A value = 1 indicates dyspnea ony for heavy efforts, A value = 2 indicates dyspnea for moderate efforts. A value = 3 indicates dyspnea for mild efforts. A value = 4 indicates dyspnea at rest.
Flow-mediated dilation (FMD); | at baseline and after 28 days of intensive pulmonary rehabilitation
  FMD evaluates the alterations of the diameter of the brachial artery in response to an induced ischemic stimulus. FMD has been widely used in clinical research and allows the studying of the influence of diseases and treatment interventions on endothelial function.
Fractional exhaled nitric oxide (FeNO) | at baseline and after 28 days of intensive pulmonary rehabilitation
  Fractional exhaled nitric oxide (FeNO) is an endogenous gaseous molecule which can be measured in human breath. Higher FeNO values have been linked airway inflammation. A cut-off of 25 parts per billion (ppb) has been suggested in order to discriminate between a normal exam (FeNO < 25 ppb) and an altered one (FeNO > or = 25 ppb).
Muscle Strength | at baseline and after 28 days of intensive pulmonary rehabilitation
  Muscle strength will be measured with a handgrip device, which consists of a handle-shaped dynamometer which is able to calculate the handgrip's strength (expressed in Newton units).

CONTACTS AND LOCATIONS:
Overall Officials: mauro maniscalco, Principal Investigator — IRCCS Maugeri Telese
Locations (3):
- Italy (3):
  - Istituti Clinici Scientifici Maugeri Irccs, Telese Terme, Benevento
  - Istituti Clinici Scientifici Maugeri IRCCS, Lumezzane, Brescia
  - Istituti Clinici Scientifici Maugeri IRCCS, Bari

IPD SHARING:
Plan to Share IPD: No